CLINICAL TRIAL: NCT06597006
Title: Two Part (Double-blind Inclisiran Versus Placebo [Year 1] Followed by Open-label Inclisiran [Year 2]) Randomized Multicenter Study to Evaluate Safety, Tolerability, and Efficacy of Inclisiran in Children (2 to Less Than 12 Years) With Homozygous Familial Hypercholesterolemia and Elevated LDL-cholesterol
Brief Title: Study to Evaluate Safety, Tolerability and Efficacy of Inclisiran in Children With Homozygous Familial Hypercholesterolemia
Acronym: ORION-19
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CKJX839C12304; 2024-514595-41 (EudraCT Number)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Familial Hypercholesterolemia - Homozygous
Keywords: Homozygous familial hypercholesterolemia (HoFH),; LDL-cholesterol (LDL-C), children, pediatric,; small interfering ribonucleic acid (siRNA),; inclisiran,; Familial Hypercholesterolemia,; Homozygous FH,; Hypercholesterolemia,; Lipoprotein(a),; Hyperlipidemia,; Dyslipidemia,; Cardiovascular Diseases,; Heart Failure,; Cholesterol,; Aortic Stenosis
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia; Hyperlipoproteinemia Type II; Hypercholesterolemia; Hyperlipidemias; Dyslipidemias; Cardiovascular Diseases; Heart Failure; Aortic Valve Stenosis | interventions — ALN-PCS; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel (Year 1) to single-group (Year 2)
Who Masked: Participant, Investigator
Masking Description: Masked (Year 1) to No Masking (Year 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inclisiran (Experimental): Year 1 - inclisiran sodium subcutaneous injection (given at Days 1, 90, and 270) Day 360 only - placebo subcutaneous injection Year 2 - inclisiran sodium subcutaneous injection (given at Days 450 and 630)
  Interventions: Drug: Inclisiran
- Placebo (Placebo Comparator): Year 1 - placebo subcutaneous injection (given at Days 1, 90 and 270) Year 2 - inclisiran sodium subcutaneous injection (given at Days 360, 450, and 630)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inclisiran — Inclisiran (inclisiran sodium 300 mg subcutaneous (s.c.) for participants with body weight ≥23 kg, inclisiran sodium 180 mg s.c. for participants with body weight <23 kg to ≥16 kg, or inclisiran sodium 100 mg s.c. for participants with body weight <16 kg. The dose level is based on the participant's body weight on Day 1 (for Part 1) and Day 360 (for Part 2), respectively.
  Other Names: KJX839
  Arms: Inclisiran
Drug: Placebo — Sterile normal saline (0.9% sodium chloride in water for subcutaneous injection)
  Other Names: saline solution
  Arms: Placebo

SUMMARY:
This is a pivotal phase III study designed to evaluate safety, tolerability, and efficacy of inclisiran in children (aged 2 to <12 years) with homozygous familial hypercholesterolemia (HoFH) and elevated low density lipoprotein cholesterol (LDLC).

DETAILED DESCRIPTION:
This is a two-part (1 year double-blind inclisiran versus placebo / 1 year open-label inclisiran) multicenter study designed to evaluate safety, tolerability, and efficacy of inclisiran in children (aged 2 to <12 years) with homozygous familial hypercholesterolemia (HoFH) and elevated low density lipoprotein cholesterol (LDL-C) on stable standard of care background lipid-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, 2 to <12 years of age at screening
* HoFH diagnosed by genetic confirmation

  - Note: Participants with known null (negative) mutations in both LDLR alleles are not eligible (see also exclusion criteria)
* Fasting LDL-C >130 mg/dL (3.4 mmol/L) at screening
* On an optimal dose of statin (investigator's discretion), unless statin intolerant, with or without other lipid-lowering therapy (e.g. ezetimibe)
* Participants on lipid-lowering therapies (such as e.g. statins, ezetimibe) must be on a stable dose for ≥30 days before screening with no planned medication or dose changes during study participation
* Participants on a documented regimen of LDL-apheresis for ≥ 3 months before screening will be allowed to continue the apheresis during the study, if needed. The apheresis schedule/settings/duration must be stable prior to screening, are not allowed to change during the double-blind period of the trial and must permit that an apheresis coincides with each study visit.

Exclusion Criteria:

* Documented evidence of a null (negative) mutation in both LDLR alleles
* Previous treatment (within 90 days of screening) with monoclonal antibodies directed towards PCSK9
* History of poor response to therapy with any monoclonal antibody directed towards PCSK9 (e.g. <15% reduction in LDL-C)
* Treatment with mipomersen or lomitapide (within 5 months of screening)
* Secondary hypercholesterolemia, e.g. hypothyroidism or nephrotic syndrome
* Heterozygous familial hypercholesterolemia (HeFH)
* Body weight (at the screening and/or randomization (Day 1) visit) <16 kg for participants 6 to <12 years (at screening) or <11 kg for participants 2 to <6 years (at screening)
* Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or unexplained alanine aminotransferase (ALT), aspartate aminotransferase (AST) elevation >3x ULN, or total bilirubin elevation >2x ULN (except patients with Gilbert's syndrome)
* Pregnant or nursing females
* Recent and/or planned use of other investigational medicinal products or devices

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2028-03-23 (Estimated); Study Completion 2029-04-15 (Estimated)

PRIMARY OUTCOMES:
Percentage change in LDL-C from baseline to Day 330 (Year 1) | Baseline and Day 330
  Evaluate the effect of inclisiran compared to placebo on reducing LDL-C [percent change] at Day 330

SECONDARY OUTCOMES:
Time-adjusted percent change in LDL-C from baseline after Day 90 and up to Day 330 (Year 1) | Baseline, after Day 90 up to Day 330
  Evaluate the effect of inclisiran compared to placebo on reducing LDL-C [time-adjusted percent change] over Year 1
Percent change in LDL-C, total cholesterol, non-HDL-C, triglycerides, HDL-C, VLDL-C from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time
Percent change in PCSK9 from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time
Percent change in Apo B, Apo A1 from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time
Absolute change in LDL-C, total cholesterol, non-HDL-C, triglycerides, HDL-C, VLDL-C from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time
Absolute change in PCSK9 from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time
Absolute change in Apo B, Apo A1 from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time
Percent change in Lp(a) from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time
Absolute change in Lp(a) from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (3):
  - UC San Francisco Medical Center, San Francisco, California
  - Childrens National Hospital, Washington D.C., District of Columbia
  - Washington Univ School Of Medicine, St Louis, Missouri
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Beijing, Beijing Municipality, China
- Novartis Investigative Site, Frankfurt am Main, Hesse, Germany
- Novartis Investigative Site, Ioannina, Greece
- Novartis Investigative Site, Kota Bharu, Kelantan, Malaysia
- Novartis Investigative Site, Amsterdam, North Holland, Netherlands
- Novartis Investigative Site, Bloemfontein, Free State, South Africa
- Taiwan (2):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Adana, Saricam
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Izmir
- Novartis Investigative Site, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.